CLINICAL TRIAL: NCT00680589
Title: Injection of AJCC Stage IIB, IIC, III and IV Melanoma Patients With Mouse Tyrp2 DNA: A Phase I Trial to Assess Safety and Immune Response
Brief Title: Patients With Mouse Tyrp2 DNA: A Phase I Trial to Assess Safety and Immune Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Jedd Wolchok, MD, Memorial Sloan-Kettering Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-052
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Melanoma
Keywords: TYRP2 DNA Vaccine
MeSH Terms: conditions — Melanoma

ARMS (1):
- 1 (Experimental): Injection of mouse TYRP2 DNA in patients with highrisk melanoma.
  Interventions: Biological: injection of mouse TYRP2 DNA

INTERVENTIONS:
Biological: injection of mouse TYRP2 DNA — Cohorts of three patients will receive injections with mouse TYRP2 DNA delivered intramuscularly at four different dose levels (500, 2000, 4000 or 8000 μg) every three weeks for six injections.

SUMMARY:
The goal of this study is to find out about the safety of injecting the gene (DNA) for mouse TYRP2 in patients with melanoma. DNA is a material that contains the information needed to produce many substances in the body. TYRP2 is a substance found in melanoma cells that helps to produce their black color. The DNA used in this study is the gene for mouse TYRP2.

The gene is introduced into bacteria, which are grown in large quantities. The DNA vaccine is then made from bacteria that is inactive.

We would like to see if we can immunize patients against TYRP2 by injecting mouse TYRP2 DNA. We will also follow the patients closely to see if there are any side effects. Mouse TYRP2 DNA is very similar to human TYRP2 DNA. We believe, based on lab experiments, that injection of mouse TYRP2 DNA could result in the production of immune substances (antibodies and T cells) that recognize melanoma cells. Antibodies are substances produced by your immune system to defend your body against bacteria and viruses. T cells are a type of white blood cell that can also fight infections. The small differences between mouse and human TYRP2 may allow your immune system to make the antibodies and T cells against melanoma. There is no evidence yet that injection of TYRP2 DNA results in any clinical benefit in patients.

ELIGIBILITY:
Inclusion Criteria:

* For all patients, pathology slides must be reviewed by the Memorial Hospital Department of Pathology for confirmation of melanoma diagnosis.
* Patients must be HLA-A*0201 positive.
* Patients must have a Karnofsky performance status of at least 80.
* Patients must be free of detectable brain metastases.
* Patients must have adequate organ and marrow function as defined below:
* WBC ≥ than or = to 3,000/μL
* Absolute neutrophil count ≥ than or = to 1,500/μL
* Platelets ≥ than or = to 100,000/μL
* Total bilirubin ≤ than or = to 1.5X upper normal institutional limits
* LDH ≤ than or = to 2 X institutional upper limit of normal
* Albumin ≥ than or = to 3.5 mg/dl
* Creatinine ≤ than or = to 2.0 mg/dl
* Hemoglobin ≥ than or = to 10 Gm/dl
* Liver AST, ALT ≤ than or = to 2.5 x ULN
* Patients must have no known HIV positivity
* Pediatric patients are eligible if weight is > 25 kg and parent/guardian completes informed assent process.
* Patients must understand and sign an informed consent and have specifically declined all standard or approved therapies for which they would be considered eligible. Parent or legal guardians of patients who are minors will sign the informed consent form.
* As part of the consent process, patients must agree to use contraception while on study.

Exclusion Criteria:

* Patients who have had chemotherapy, immunotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. For nitrosoureas, at last six weeks must have elapsed.
* Patients with Grade I fever, active infection, or antibiotics within 72 hours prior to study.
* Patients who have previously been immunized with any class of vaccine containing TYRP2, including whole cell, shed antigen or cell lysate vaccine.
* Patients with a history of collagen vascular, rheumatological, or other autoimmune disorders.
* Any medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to respond immunologically to vaccines is grounds for exclusion, at the discretion of the Principal Investigator or co-Principal Investigators.
* Patients who have preexisting retinal or choroidal eye disease.
* Patients with serious underlying medical conditions that could be exacerbated by participation, active infections requiring antimicrobial drugs or active bleeding.
* Pregnant women or women who are nursing are not eligible. Women of child-bearing potential and sexually active men must be using appropriate contraception during the course of this study. Women of child-bearing potential must not be pregnant (negative βHCG within 2 weeks of immunization) nor be nursing during treatment.
* Patients receiving other investigational agents.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and feasibility of intra-muscular DNA injection with mouse TYRP2 DNA. Doses will be escalated by groups to determine the maximal tolerated dose. | conclusion of study

SECONDARY OUTCOMES:
A secondary endpoint is to observe the patients for evidence of any antitumor response generated after immunizations. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Jedd Wolchok, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org